CLINICAL TRIAL: NCT01475019
Title: The Effect of Weight Loss With Orlistat or Sibutramine Administration , Hypocaloric Diet and Physical Exercise , on AMH Levels, in Women With Polycystic Ovary Syndrome
Brief Title: The Effect of Weight Loss on Anti-Müllerian Hormone Levels in Women With Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, C.VOSNAKIS, Obstetrician- Gynecologist, Scientific Assosiate of Medical School of Aristotle University, Thessaloniki, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A1732,2011
Record Dates: First submitted 2011-11-14; First posted 2011-11-21 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Obesity; Polycystic Ovaries Syndrome
Keywords: Obesity; Polycystic Ovaries Syndrome; Orlistat; Sibutramine; Androgen levels; Insulin resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Orlistat; sibutramine; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PCOS obese Orlistat (Experimental): Obese PCOS women treated with Orlistat, diet and physical exercise
  Interventions: Drug: Orlistat
- Obese Orlistat (Experimental): Obese women (non PCOS) treated with Orlistat, diet and physical exercise
  Interventions: Drug: Orlistat
- PCOS obese diet (Experimental): Obese PCOS women treated with diet and physical exercise
  Interventions: Behavioral: Diet and physical exercise
- PCOS obese Sibutramine (Experimental): Obese PCOS women treated with Sibutramine, diet and physical exercise
  Interventions: Drug: Sibutramine

INTERVENTIONS:
Drug: Orlistat — Tablet, 120 mg, three times daily, for six months
  Arms: Obese Orlistat; PCOS obese Orlistat
Drug: Sibutramine — Tablet, 10 mg, once daily, for six months
  Arms: PCOS obese Sibutramine
Behavioral: Diet and physical exercise — Hypocaloric diet and regular physical exercise
  Arms: PCOS obese diet

SUMMARY:
The first aim of the investigators study, was to investigate the combined effect of diet,physical exercise and orlistat, for 24 weeks, on serum Anti-Müllerian Hormone (AMH) levels in obese women with polycystic ovary syndrome (PCOS) and in obese controls.

The other aim of the investigators study, was to examine the effect of hypocaloric diet,physical exercise plus sibutramine on serum AMH levels, body composition, hormonal and metabolic parameters in overweight and obese patients with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
The first aim of our study, was to investigate the combined effect of diet,physical exercise and orlistat, for 24 weeks, on serum Anti-Müllerian Hormone (AMH) levels in obese women with polycystic ovary syndrome (PCOS) and in obese controls.

The study included sixty one (61) women with PCOS (mean age: 26.11±6.86 and mean body mass index: 34.83±6.39), matched for age and body mass index (BMI) with twenty (20) obese women without PCOS (mean age: 26.95±4.77 and mean BMI: 36.79±6.98). Diagnosis of PCOS was based on the 2003 Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus criteria.

Briefly, a moderate daily physical activity and a normal-protein, energy restricted diet were prescribed based on a calculated individual basal metabolic rate (BMR) of all women (BMR-600 kcal/d), for a period of 24 weeks. In addition, orlistat (Xenical, Roche S.A., Greece; 120 mg, 3 times per day) was administered before each meal, for 24 weeks. At baseline, week 12, and week 24, at 9:00 AM, after an overnight fast, subjects were weighed. Waist and hip circumferences were measured in duplicate. Blood samples were collected and the basal serum levels of AMH, FSH, LH, PRL, T, D4A, DHEAS, 17a-hydroxyprogesterone (17a-OHP), SHBG, glucose, and insulin were measured. AMH concentrations were measured with an enzymatically amplified two-sided immunoassay [DSL-10-14400 Active Müllerian Inhibiting Substance/AMH enzyme-linked immunosorbent assay (ELISA) kit, DSL Laboratories, Webster, TX]. The theoretical sensitivity of the method is 0.006 ng/ml, the intra-assay coefficient of variation for high values is 3.3% and the interassay coefficient of variation for high values is 6.7%.

We also studied the changes of mean number of follicles (expressed as the mean number of follicles of both ovaries= follicles of right ovary+ follicles of left ovary/2) and mean ovarian volume (expressed as the mean volume of both ovaries= volume of right ovary+ volume of left ovary/2).

The other aim of our study, was to examine the effect of hypocaloric diet,physical exercise plus sibutramine on serum AMH levels, body composition, hormonal and metabolic parameters in overweight and obese patients with polycystic ovary syndrome (PCOS).

Outpatients, premenopausal, nonpregnant, nonlactating, overweight and obese women (body mass index, BMI >27), 18 years of age and older with PCOS were recruited for this study. The study included fifty seven (57) women with PCOS (mean age: 26.11±6.86 and mean body mass index: 34.83±6.39) who, besides diet and exercise, received Sibutramine treatment, matched for age and body mass index (BMI) with nineteen (19) obese women with PCOS (mean age: 26.95±4.77 and mean BMI: 36.79±6.98) treated only with diet and exercise. Diagnosis of PCOS was based on the 2003 Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus criteria . Women with no classical 21-hydroxylase deficiency, hyperprolactinemia, adrenal or ovarian tumor and Cushing's disease were excluded by the appropriate tests. Other exclusion criteria were hypertension, thyroid dysfunction, overt diabetes mellitus and concomitant treatment, such as antihypertensive drugs, selective serotonin reuptake inhibitor or other SNRI drug, oral contraceptive pills or any other antiandrogen treatment (cyproterone acetate, spirolactone, luteinizing hormone (LH) release hormone agonist) and insulin-sensitizing agents (metformin, pioglitazone, rosiglitazone) that may interact with insulin sensitivity and lipid profile.

Briefly, all patients were placed in a hypocaloric diet plus sibutramine (10mg per day) for the first month and then on a hypocaloric diet plus sibutramine (10mg per day) or hypocaloric diet only for the subsequent 6 months. A moderate physical activity (3 hours per week) and a normal-protein, energy restricted diet were prescribed based on a calculated individual basal metabolic rate (BMR) of all women (BMR-600 kcal/d), for a period of 24 weeks.

At baseline, week 12, and week 24, at 9:00 AM, after an overnight fast, subjects were weighed. Waist and hip circumferences were measured in duplicate. Blood samples were collected and the basal serum levels of AMH, FSH, LH, PRL, T, D4A, DHEAS, 17a-hydroxyprogesterone (17a-OHP), SHBG, glucose, and insulin were measured. AMH concentrations were measured with an enzymatically amplified two-sided immunoassay [DSL-10-14400 Active Müllerian Inhibiting Substance/AMH enzyme-linked immunosorbent assay (ELISA) kit, DSL Laboratories, Webster, TX].

ELIGIBILITY:
Inclusion Criteria:

* premenopausal,
* nonpregnant,
* nonlactating,
* overweight and obese women

Exclusion Criteria:

* classical 21-hydroxylase deficiency,
* hyperprolactinemia,
* adrenal or ovarian tumor and Cushing's disease

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-01; Primary Completion 2010-01 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Anti- Mullerian hormone (AMH) levels | 6 months

SECONDARY OUTCOMES:
Weight loss | 6 months
Androgen levels | 6 months
  Free androgen index, Testosterone, 17OH Progesterone, D4 Andostenedione, Testosterone to Androstenedione ratio
Follicular number | 6 months
  Mean follicular number
Gonadotrophins | 6 months
  Follicular Stimulating Hormone (FSH), Luteneizing Hormone (LH), LH to FSH ratio

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Panidis, PhD, Study Director — Aristotle University of Thessaloniki Medical School
Locations (1):
- Aristotle University of Thessaloniki Medical School, Thessaloniki, Thessaloniki, Greece